CLINICAL TRIAL: NCT02728024
Title: Assessing Psychosocial and Supportive Care Needs in Patients With Gliomas
Acronym: ERASMUS
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Ulm (Other); Klinikum Stuttgart (Other)
Responsible Party: Principal Investigator, Dr. med. Mirjam Renovanz, MD, Johannes Gutenberg University Mainz
Other Study IDs: ERASMUS
Record Dates: First submitted 2016-03-22; First posted 2016-04-05 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Complete the questionnaires with personal aid
  Interventions: Other: Missing items, Errors in Completion, Difficulties
- B: questionnaires are completed by patients alone
  Interventions: Other: Missing items, Errors in Completion, Difficulties

INTERVENTIONS:
Other: Missing items, Errors in Completion, Difficulties

SUMMARY:
The study is undertaken at three German neurosurgical centers (Ulm, Mainz, Stuttgart) between March 2014 and March 2015. Inclusion criteria were age ≥ 18 and ≤ 80, diagnosis of glioma WHO° II-IV, absence of aphasia impairing communication or consent. In an outpatient setting all eligible patients with gliomas were screened for distress (Distress Thermometer (DT)) and their need for psychosocial support (Supportive Care Needs Survey-SF34-G (SCNS)). Simultaneously their HRQoL was assessed (EORTC QLQ-C30+BN-20 Vers. 3).

Patients at different disease stages were asked to fill out the questionnaires. At two study centers patients were asked to complete the questionnaires prior to their appointment with personal instructions in randomly selected cases. At the third study center, they completed the questionnaires after their outpatient appointment with personal aid and instructions. At the time of investigation, patients were at different stages of treatment (chemotherapy, radiation, re-chemotherapy, re-radiation, none, etc.).

DETAILED DESCRIPTION:
Study design

In three neuro-oncological outpatient departments of the three study centers (two of them are university medical centers, one a teaching hospital), glioma patients were assessed between March 2014 and March 2015 using three questionnaires. Due to the infrastructure of the outpatient departments, assessing ment of supportive care needs, HRQoL, and distress, by the questionnaires was performed either with the opportunity of personal support by the study members (group A) or by patients alone (group B).

In group A, a member of the study group (no caregivers) offered help and stayed with the patient the whole time while the patient was filling in the questionnaires. Every patient received an explanation and was offered additional support. If questions occurred or the patient was not able to fill in the questionnaires by him-/herself, the study member helped by answering questions, assisting or describing the questionnaires in detail or even reading out the questions to the patient and filling in the answers which were chosen by the patient. The extent of the assistance by the study members varied depending on the impairment of the patient. Occurrence and details of difficulties in completion were assessed by a feedback form especially developed for this study which was filled in by the member of the study group after completing the instruments. If patients were unable to complete the questionnaires by themselves, the reason for this was documented by the interviewer (e.g. neurocognitive impairment, physical disability, decreased attention span, etc. based and categorized on clinical judgement of the interviewer).

In group B, patients completed the questionnaires on their own. In one study center, Allocation to study groups was randomized in one study center (block randomization independently provided by Institute of Medical Biostatistics, Mainz). Patients in the other two centers were either always group A or always group B.

Furthermore, socio-demographic data, tumor stage, Karnofsky Performance Status (KPS), pre-and postsurgical clinical characteristics (e.g. postoperative tumor remnant, localization of the tumor), and adjuvant therapies were documented.

The study was undertaken in concordance with national law, institutional ethical standards and the Helsinki Declaration, and the ethic commissions of all three study centers approved the study.

Patient population

Selection criteria for this study were:

1. a glial cerebral tumor (astrocytoma, oligoastrocytoma, oligodendroglioma, glioblastoma), as diagnosed by the local neuro- pathologist in the study center;
2. patient is affiliated with the neuro-oncological outpatient center in one of the three study centers;
3. patient is able to understand and respond to the questions;
4. informed consent of the patient.

PRO Questionnaires

For the first assessment, the SCNS-SF34-G, Distress Thermometer (DT), EORTC -QLQ- C30 + EORTC QLQ-BN20 and were used, for the second assessment after 3-5 months the SCNS-ST9, DT, and EORTC-QLQ-C30 + EORTC QLQ-BN-20 were used.

The SCNS-SF34, a short-form version of the SCNS long-form, is a self-reporting instrument measuring patients' needs of supportive care. It consists of five domains: health system and information, psychological, physical and daily living, patient care and support, and sexuality needs. Lehmann et al. demonstrated adequate psychometric properties in the German version. On a 5-point Likert scale, patients indicate if they are in need of support and, if so, the extent of their need (1 = no need, not applicable; 2 = no need, satisfied; 3 = low need; 4 = moderate need; 5 = high need).

The SCNS-SF9 is an ultrashort screening instrument developed of the SCNS-SF34 consisting of nine questions. The structure of the screening instruments is similar to the SCNS-SF34-G with the same 5-point Likert scale as described.

The EORTC QLQ-C30 is a frequently used questionnaire including 30 items to assess quality of life in oncological patients and includes five functional scores (physical, role, emotional, social, and cognitive function). The reliability and validity of the instrument have been approved in many clinical trials, and it has been translated into 85 languages. The brain module (QLQ-BN20) comprises 20 questions developed for brain tumor patients and includes four functional scales.

The Distress Thermometer (DT), a self-reporting instrument, evaluates psychological distress using a visual analogue scale along with 40 items assessing financial, physical, emotional and spiritual concerns (problem list). Developed by the National Comprehensive Cancer Network (NCCN), the German version was adapted in 2007. A score of six or above on the visual analogue scale is recommended as a cut-off for a clinically significant level of distress for brain tumor patients. The DT is well accepted for in oncological patients.

Endpoints

The primary evaluation of feasibility of the questionnaires in clinical routine was analyzed by analyzing the occurrence of missing values and the occurrence of errors in the SCNS-SF34-G and SCNS-ST9. Missing values were assessed in the categories single missing items (at least one item per questionnaire missing) and missing questionnaire (complete questionnaire was not filled in). An error was defined as multiple responses for an item where only one response per patient would have been correct. For both outcomes comparisons were made to the EORTC QLQ-C30+BN20 and DT as well as between groups A and B.

The study members providing support for the patients of group A gave feasibility feedback regarding the difficulties occurred during the assessment after each patient using a 10-item feedback form developed for this study with the following items:

* Occurrence of difficulties (yes/no)
* Time needed for assessment (10-20min, 21-30min, 31-40min, 41-50 min, >51min)
* Impairment of the patients (none, cognitive, psychological, physical)
* If problems during the assessment occurred (none/rare/moderate/severe; defined by the frequency of questions asked by the patients)
* Which difficulties occurred (understanding questionnaire/complexity of questionnaire/extend of questions/physical problems e.g. paresis)
* Which questionnaire caused problems (EORTC/DT/SCNS)
* Which questionnaires were filled in with/without assistance
* Aid intensity level provided by the study members (assistance in one, two or all three questionnaires).

Where possible these items were also analyzed in comparison to the other PRO instruments.

Difficulties occurred in the SCNS were compared to the EORTC QLQ-C30+BN20 and DT whenever possible.

ELIGIBILITY:
Inclusion criteria:

* Harboring a glial cerebral tumor (astrocytoma, oligoastrocytoma, oligodendroglioma, glioblastoma), as diagnosed by the local neuro- pathologist in the study Center
* Patient is affiliated with the neuro-oncological outpatient center in one of the three study Centers
* Patient is able to understand and respond to the questions
* Informed consent of the Patient
* Age >18, <80 years

Exclusion criteria:

* Absence of inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selection criteria for this study were 1) a glial cerebral tumor (astrocytoma, oligoastrocytoma, oligodendroglioma, glioblastoma), as diagnosed by the local neuro- pathologist in the study center; 2) patient is affiliated with the neuro-oncological outpatient center in one of the three study centers; 3) patient is able to understand and respond to the questions; 4) informed consent of the patient.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of missing items in questionnaires | Baseline
  Number of missing items per questionnaire

SECONDARY OUTCOMES:
Definition of discrimination thresholds for glioma patients with and without distress based bon EORTC QLQ-C30 functioning scores. | Baseline
  Unitless PRO measures of SCNS-SF34-G were grouped into categories corresponding to the functioning scales, HRQoL scale and selected symptom scales of the EORTC QLQ-C30/BN20: physical function (physf), role function (rolef), emotional function (emof), cognitive function (cognf), social function (socf), quality of life (GHS), future uncertainty (FU), fatigue, and motor dysfunction). SCNS scores >3 were defined as need for supportive care with the respective issue. Decision thresholds for the corresponding EORTC QLQ functioning scores were determined using receiver operating characteristics.
Definition of discrimination thresholds for glioma patients with and without supportive care needs based on EORTC QLQ-C30 functioning scores. | Baseline
  Items of the problem list of the DT questionnaire were grouped into categories corresponding to the functioning scales, HRQoL scale and selected symptom scales of the EORTC QLQ-C30/BN20: physical function (physf), role function (rolef), emotional function (emof), cognitive function (cognf), social function (socf), quality of life (GHS), future uncertainty (FU), fatigue, and motor dysfunction). Decision thresholds for the corresponding EORTC QLQ functioning scores were determined using receiver operating characteristics. DT >6 was defined significant distress.

IPD SHARING:
Plan to Share IPD: No